CLINICAL TRIAL: NCT07183072
Title: Investigating the Relationship Between the Biopsychosocial Status of Individuals Diagnosed With Scleroderma and Their Physical Performance and Functionality
Brief Title: Patients Diagnosed With Scleroderma: Physical Performance and Functionality
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Orkun Tüfekçi, Principal Investigator, PT, PhD(c), Hacettepe University
Other Study IDs: SBA 25/529
Record Dates: First submitted 2025-09-13; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-08

CONDITIONS: Systemic Sclerosis (SSc); Scleroderma; Scleroderma (Limited and Diffuse); Scleroderma, Localized; Functionality
Keywords: Juvenile scleroderma; scleroderma; systemic sclerosis; physical performance; functionality
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse; Scleroderma, Localized; Juvenile-onset scleroderma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases diagnosed with scleroderma: Child and adult scleroderma patients who visited the rheumatology outpatient clinic at a university hospital will complete a questionnaire.
  Interventions: Other: Questionnaire and functionality application for child and adult scleroderma patients

INTERVENTIONS:
Other: Questionnaire and functionality application for child and adult scleroderma patients — Scales and functionality tests will be applied to cases diagnosed with scleroderma

SUMMARY:
Physical functionality and performance are important for individuals diagnosed with scleroderma. There is a need to address children and adults diagnosed with scleroderma comprehensively and to evaluate them on a biopsychosocial basis to support their disease management. In light of all this literature, the aim was to evaluate the biopsychosocial characteristics of both pediatric and adult scleroderma patients and to examine their physical performance and functionality.

Additionally, this study aims to identify effective tests that can be used in future research to assess physical performance and functionality in individuals diagnosed with scleroderma.

ELIGIBILITY:
*For a child diagnosed with scleroderma*

Inclusion Criteria:

* Cases diagnosed with scleroderma,
* Cases aged 7-18 years will be included.

Exclusion Criteria:

* Advanced heart/lung/liver/kidney disease, neurological disease, and malignancies
* Cases that are not willing to participate in the study will be excluded.
* Having participated in a regular exercise program for the past 3 months
* Individuals who are not willing to participate in the study

*For adults diagnosed with scleroderma*

Inclusion Criteria:

* Individuals diagnosed with scleroderma,
* Individuals over the age of 18 will be included.

Exclusion Criteria:

* Advanced heart/lung/liver/kidney disease, neurological disease, and malignancies
* Individuals who are not willing to participate in the study will be excluded.
* Having participated in a regular exercise program for the past 3 months
* Individuals who are not willing to participate in the study

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of individuals who come to the university hospital for routine controls.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08-04 (Estimated)

PRIMARY OUTCOMES:
6-Minute Walk Test | Two weeks
  Participants are asked to walk as quickly as they can along a 30-meter corridor. The total distance will be measured in meters. Fatigue, pain and dyspnea will be monitored using the Modified Borg Scale.
Timed Up and Go Test | Two weeks
  The time it takes for a person to get up from a chair with back support, walk 3 meters at a normal pace, and return to the chair is measured in seconds to evaluate lower extremity balance. The test will be performed 3 times.
10-Step Stair Climbing Test | Two weeks
  To assess the subject's lower extremity strength and dynamic balance, the time taken to quickly climb and descend a staircase with 10 steps, each measuring 16-20 cm high and equipped with a handrail, is recorded in seconds. The test is repeated three times, and the times are recorded.
10-meter walk test | Two weeks
  The individual is on a 10-meter path. The assessment is performed in three repetitions and recorded in seconds.
30-second sit-to-stand test | Two weeks
  It is performed to evaluate lower extremity endurance by having the individual stand up from a chair with their arms crossed over their chest and then sit back down. The individual is instructed to repeat this as quickly as possible for 30 seconds. The score for this assessment is the number of times the person fully stands up from a sitting position with arms crossed within 30 seconds.
Glittre Activities of Daily Living Test | Two weeks
  It consists of a cycle of standardized activities such as walking, carrying weights, climbing stairs, and moving objects on a shelf. The equipment required for the test includes a chair, steps, a shelf, a backpack, weights (0.5 kg-2.5 kg), and a stopwatch. The patient completes the 10-meter course created for the test for five laps, and the time is recorded.

SECONDARY OUTCOMES:
Childhood Health Assessment Questionnaire (CHAQ) | Two weeks
  It assesses the functional abilities of children diagnosed with rheumatic diseases in their daily living activities. It consists of eight subscales (dressing and personal care, standing up, eating, walking, body care, reaching, grasping, activities) (0-3) and also assesses pain and general well-being using a visual analog scale (0-100). A high score indicates low functionality.
Juvenile Arthritis Quality of Life Questionnaire (JAQQ) | Two weeks
  It consists of 74 items covering various health domains, including physical functioning, emotional well-being, and general symptoms. The items are divided into four dimensions related to the child's quality of life: gross motor function (GMF), fine motor function (FMF), psychosocial function (PF), and systemic or general symptoms (SGS). Each domain is scored on a Likert-type scale from 1 to 7; higher scores indicate poorer health-related quality of life. There is also a "not applicable to me" option for the items. The scale also includes a pain measurement (10 cm Visual Analog Scale (VAS)) to assess pain, but this score is not included in the total score.
Juvenile Arthritis Biopsychosocial Scale-JAB-Q-Patient | Two weeks
  It is a patient/parent-centered measurement method that helps assess the patient's biopsychosocial aspects, such as disease activity, posture, functional and psychosocial status, fatigue, and school performance. The results from the questions are used to assess the functional status of children, while their psychosocial status is recorded based on their answers to 21 questions (ranging from 0 to 358). A high score indicates a poor psychosocial status.
Juvenile Arthritis Biopsychosocial Scale-JAB-Q-Family | Two weeks
  JAB-Q is a multidimensional questionnaire and a parent (family) form. Developed in Turkish by Ünal and colleagues, the questionnaire is completed by one of the child's parents. The family form evaluates the parents' biopsychosocial status from their own perspective and provides scores ranging from 0 to 102. Higher scores indicate a worse biopsychosocial status.
Pain Catastrophizing Scale-Parent (PCS-P) | Two weeks
  It is assessed using a 5-point Likert scale ranging from 0 (never) to 4 (always) and consists of 13 items. Similar to the child questionnaire, it assesses 3 domains: rumination, magnification, and helplessness. A total score between 0 and 52 is obtained; higher scores reflect a higher level of catastrophizing in parents.
Child and Adolescent Scale of Participation (CASP) | Two weeks
  It is a 20-question survey that evaluates the community participation of children and adolescents in school, neighborhood, and local settings. The survey is divided into four sections: 6 questions about home participation, four questions on neighborhood and community involvement, five questions regarding school participation, and five questions on home and community engagement. It is rated on a scale of "expected for their age (full participation), somewhat limited, very limited, unable to participate, and inapplicable." The survey is completed by the child's family or primary caregiver. The person filling out the questionnaire is asked to select the answer that best describes the child's level of participation. The assessment is scored out of 100 points, with higher scores reflecting a greater level of participation.
Scleroderma Health Assessment Questionnaire (SHAQ) | Two weeks
  It was developed by adding five questions to the HAQ regarding Raynaud's phenomenon, digital ulcers, gastrointestinal, pulmonary, and general scleroderma symptoms, to be rated on a 15 cm line. The SHAQ total score ranges from 0 to 3. A high score indicates low functionality.
Cognitive Exercise Therapy Approach-Biopsychosocial Questionnaire (BETY-BQ) | Two weeks
  It was standardized as a biopsychosocial assessment tool and is scored using a 5-point Likert scale, with each item rated from 0 to 4 points. A high total score on the 30-item scale indicates a high level of biopsychosocial impact.
Short Form-36 (SF-36) | Two weeks
  It will be used to determine an individual's quality of life levels. Each sub-parameter is scored between 0 and 100 points, with a high score indicating good health status. The SF-36 scale has eight sub-parameters: general health perception, physical function, social function, pain, mental health, role difficulty due to physical reasons, role difficulty due to emotional reasons, and vitality. It contains 11 questions consisting of a total of 36 items.
Central Sensitization Scale (CSS) | Two weeks
  It is a 40-item scale, scored on a 0-4 Likert scale, that assesses symptoms related to central sensitization. A score above 40 is interpreted as an indicator of central sensitization.
Hospital Anxiety and Depression Scale (HADS) | Two weeks
  It consists of fourteen questions, with odd-numbered questions assessing anxiety and even-numbered questions assessing depression. The options are scored from 0 to 3, with higher scores indicating a worse emotional state. The Turkish cut-off values for the scale are 10 for the anxiety subscale and 7 for the depression subscale.
Modified Rodnan skin score (MRSS) | Two weeks
  A pediatric and adult rheumatologist assessed it. The MRSS evaluates skin thickening in 17 body regions, graded from 0 (normal) to 3 (severe skin thickening). The total score ranges from 0 to 51, with increased scores indicating poor skin involvement.
Localized Scleroderma Assessment Tool (LoSCAT) | Two weeks
  LoSCAT consists of two sections: the modified Localized Skin Severity Index, which measures disease activity, and the Localized Scleroderma Damage Index, which assesses damage (usually scored between 0 and 3). The Localized Skin Severity Index evaluates the color of the lesion border for erythema, skin thickness, and the presence of new lesions or lesion extension. In the Localized Scleroderma Damage Index, three areas of cutaneous damage are combined to obtain a score. These areas evaluate hyperpigmentation or hypopigmentation, whichever is more prominent, as well as dermal atrophy, subcutaneous atrophy, and dyspigmentation.
Modified Hand Mobility in Scleroderma Test (mHAMIS) | Two weeks
  It is a functional test developed specifically for scleroderma to assess an individual's hand function. It evaluates four specific hand movements (finger flexion, finger extension, finger abduction, and dorsal extension). Scores range from 0 (normal) to 3 (complete failure) for each movement, with a total score ranging from 0 to 12.
Pain Catastrophizing Scale-Children (PCS-C) | Two weeks
  It consists of 13 items that describe the different thoughts and feelings children may experience when they feel pain. The questionnaire assesses three areas: rumination, magnification, and helplessness. All items are rated on a scale from 0 (never) to 4 (always). Higher scores reflect more catastrophic beliefs about pain. The total score can range from 0 to 48.
Transition Readiness Assessment Questionnaire (TRAQ) | Two weeks
  It includes 20 items divided into five subscales. These subscales are related to "Management of Treatment" (the first four items), "Scheduling Appointments" (items 5-11), "Monitoring Health Issues" (items 12-15), "Communication with Healthcare Personnel" (items 16-17), and "Management of Daily Activities" (items 18-20). The scale uses a 5-point Likert-type scale and has a total score range of 20 to 100. The scale score reflects the level of readiness for transitioning to adult care.
Pain Catastrophizing Scale | Two weeks
  It includes 13 items that describe different thoughts and feelings that may occur when pain is experienced. The questionnaire assesses three areas: rumination, magnification, and helplessness. All items are rated on a scale from 0 (never) to 4 (always). Higher scores indicate more catastrophic pain beliefs. The total score ranges from 0 to 52.
Clinical Frailty Scale | Two weeks
  It assesses elements such as comorbidity, cognitive impairment, and disability. Frailty scores range from 1 to 9, with one meaning 'very fit' and nine meaning 'terminally ill'. A score of 5 or above is considered a sign of frailty.
Frailty Scale | Two weeks
  FRAIL is a 5-item scale developed by Morley and colleagues to evaluate frailty. Each question is scored as 0 or 1 point. The total score ranges from 0 to 5 points (0 points = Fit, 1-2 points = Pre-frail, 3-5 points = Frail).

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No